CLINICAL TRIAL: NCT00342953
Title: Extended Mortality Follow-Up of Women With Augmentation Mammoplasty
Brief Title: Study of Health Effects of Cosmetic Breast Augmentation
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903082; 03-C-N082
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Brain Cancer; Breast Cancer; Lung Cancer; Suicide
Keywords: saline; silicone; Breast Implants; augmentation mammoplasty; visk
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Lung Neoplasms; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort: Women receiving implants and other plastic surgery.

SUMMARY:
This study will examine long-term health effects of cosmetic breast augmentation (enlargement) with silicone gel breast implants. There has been concern for some time about the possible effects of breast implants on the immune system particularly regarding the development of certain connective tissue disorders and on the possibility that implants may interfere with the ability to detect breast cancers. More recently, concerns have been raised regarding the possible cancer-causing effect of the implants themselves. These concerns were heightened by reports that the polyurethane foam coating that envelops the silicone gel in some implants may dissolve and produce a chemical called 2,4,-diamino toluene (TDA), which has been linked to an increased risk of breast and other cancers in rats and mice.

To address this issue, this study will gather information from the medical records and a questionnaire survey of approximately 12,000 breast implant patients. The questionnaire will request information on perceived complications of the implants; history of breast examinations and mammograms; frequency of breast self examination; development of diseases (particularly cancers and connective tissue disorders) developed subsequent to the augmentation surgery; potential risk factors for these diseases, such as age at menarche (onset of menstruation), age at first birth, age and type of menopause (natural or due to surgery); history of breast biopsies; immune system and connective tissue disorders; cigarette smoking; alcohol consumption; family medical history, and so forth. To evaluate the results, the information will be compared with the same data on 4,000 women who underwent other plastic surgery procedures, such as rhinoplasty, facelift, liposuction, dermabrasion, eyelifts, and others, from the same practices as the breast augmentation patients.

Participants will be recruited for the study from several large reconstructive and plastic surgery practices. Among the breast implant patients, women who have had bilateral breast implants for cosmetic purposes only, and not as breast reconstruction after breast cancer surgery, will be eligible. Women with a history of breast cancer may not participate.

DETAILED DESCRIPTION:
Although approximately 2 million women in this country have undergone augmentation mammoplasty, little is known about long-term effects. There has been concern for some time regarding possible effects of implanted material on the immune system. In addition, there has been a long-standing concern that breast implants may deter the detection of breast cancers. More recently, concern has developed over the possible carcinogenicity of the material used in implants themselves. Of particular concern is the recognition that a polyurethane foam coating used to contain silicone gel in some implants is comprised of the chemicaI 2, 4-diamino toluene, or TDA, which has been linked to increased risks of breast as well as other cancers in rats and mice. To address these concerns, a retrospective cohort study of approximately 12,000 breast implant patients is proposed. It is anticipated that these women will be recruited from a number of large reconstructive and plastic surgery practices in several diverse areas. The cohort will be constructed in such a manner that a variety of different implant types are represented and an average of 10 years of follow-up on the patients is achieved. Records at the collaborating practices will be reviewed to obtain identifiers of potential study subjects, particulars of the surgery and possible co-variates for subsequent diseases. Using a variety of sources, the subjects were traced for current vital status and residence. A questionnaire will be developed and sent to the study subjects. This questionnaire will request information from the subjects on perceived complications of the implant, history of breast examinations and mammograms, frequency of breast self examinations, development of diseases subsequent to the operation (with particular interest on cancer and connective tissue disorders), and potential risk factors for the diseases of interest (e.g., age at menarche, age at first birth, age and type of menopause, family medical history, immune alterations). Because of difficulties in comparing this population to an external standard, an internal comparison cohort was also assembled. This will consist of approximately 4,000 women receiving operations from the same plastic surgery practices as the breast augmentation patients. This comparison group will consist of women undergoing a variety of cosmetic plastic surgery procedures, such as rhinoplasty. Attempts will be made to assemble a cohort with similar ages and operations dates as the breast implant patients. Records of these patients will be abstracted and follow-up pursued in the same manner as for the mammoplasty patients. The cancer incidence and mortality experience of the augmentation mammoplasty patients was compared to both general population rates (using SEER cancer incidence and U.S. mortality rates) and to that of the experience of the other plastic surgery patients. Analyses of the risk of connective tissue disorders focused solely on the internal comparisons, given the absence of available population incidence rates for these disorders. Analyses included efforts to assess risks by various implant characteristics, including age at, calendar time of, and interval since implantation. Internal analyses enabled adjustment for recognized risk factors, particularly for the cancers of interest.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

The following criteria for inclusion in the study cohort will apply:

1. Age. No age restrictions apply; patients receiving cosmetic implants at any age will be eligible for study.
2. Cosmetic augmentation only. Patients with breast reduction surgery or reconstructive surgery following breast cancer will not be included.
3. Females only. Implants in conjunction with sex change surgery will not be included.
4. Bilateral implants only. Patients with unilateral implants will not be included.
5. First occurrence of a breast implant. Patients with a previous breast implant will not be included.
6. Patients with a history of plastic surgery involving silicone exposure will not be included.
7. Patients with a history of breast cancer at or before the time of implant will not be included.
8. Patients residing in defined geographic areas at the time that their plastic surgery was sought (these areas will need to be individually defined for each study site).
9. Patients with a history of breast surgery for non-cancerous events, those with a history of cancer of sites other than the breast, and those with documented histories of connective tissue disorders will continue to be eligible for cohort inclusion, although information on these conditions will be abstracted so that separate analyses can be pursued.

For the comparison cohort, items a, c, f, g, h and i will apply. Patients currently receiving an operation involving implantation of silicon will not be included in the comparison cohort.

Ages: 21 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 13,488 women receiving cosmetic implants and 3,936 patients who had other types of plastic surgery at 18 plastic surgery practices during the period 1960-1988.
Sampling Method: Non-Probability Sample
Enrollment: 17424 (Actual)
Dates: Start 2003-01-10 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
No intervention | Indefinite
  Assessing effect of augmentative breast surgery upon breast cancer risk.

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Hoover, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baldwin CM Jr, Kaplan EN. Silicone-induced human adjuvant disease? Ann Plast Surg. 1983 Apr;10(4):270-3. doi: 10.1097/00000637-198304000-00002. PMID 6847084
- [Background] Benavent WJ. Treatment of bilateral breast carcinomas in a patient with silicone-gel breast implants. Case report. Plast Reconstr Surg. 1973 May;51(5):588-9. doi: 10.1097/00006534-197305000-00026. No abstract available. PMID 4349607
- [Background] Ashley FL. A new type of breast prosthesis. Preliminary report. Plast Reconstr Surg. 1970 May;45(5):421-4. doi: 10.1097/00006534-197005000-00001. No abstract available. PMID 5438186